CLINICAL TRIAL: NCT06964048
Title: Evaluation of Cold Plasma in Wound Healing: A Randomized Controlled Pilot Study on Chronic Venous Leg Ulcers and Diabetic Foot Ulcers.
Brief Title: Evaluation of Cold Plasma in Chronic Wound Healing
Acronym: PLASANAGENESIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Plasana Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC202401
Record Dates: First submitted 2025-04-15; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Chronic Wounds; Venous Leg Ulcer (VLU); Diabetic Foot Ulcer (DFU); Pressure Ulcer (PU)
Keywords: Chronic wounds; Venous Leg Ulcer; VLU; Diabetic Foot Ulcer; DFU; Pressure Ulcer; PU; Cold Atmospheric Plasma; CAP; Plasma; Cold Plasma; Healing; Wound Closure
MeSH Terms: conditions — Varicose Ulcer; Diabetic Foot; Pressure Ulcer | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Participants in the control group will receive the standard of care alone.
- Intervention Arm (Experimental): Participants in the intervention group will be treated according to the same protocol as the control group, with the addition of cold plasma therapy with Plasana One®, as an add-on to the standard of care.
  Interventions: Device: Cold Atmospheric Plasma treatment

INTERVENTIONS:
Device: Cold Atmospheric Plasma treatment — Participants in the intervention group will be treated with cold plasma therapy with Plasana One®, as an add-on to the standard of care.
  Other Names: CAP treatment; Plasma treatment; Plasma application; CAP application; Cold plasma therapy
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of cold atmospheric plasma treatment in promoting the healing of chronic wounds in adult participants suffering from chronic wounds. The main questions is the following: Does the application of cold atmospheric plasma accelerate wound healing compared to standard wound care alone?

Researchers will compare standard of care plus plasma treatment with standard of care alone to see if the plasma-treated group shows faster wound healing.

Participants will:

* Receive either standard wound care alone or standard wound care combined with cold atmospheric plasma treatment, depending on randomization.
* Attend scheduled hospital visits for wound care, treatment administration, and clinical assessments, including wound photography and quality of life questionnaires.
* Be followed up at home by nurses for wound care, treatment administration and clinical assessment too.
* Complete a wound-related quality of life questionnaire at baseline, at week 6, and at the end of the study.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled clinical trial evaluating the efficacy and safety of cold atmospheric plasma (CAP) therapy using the Plasana One® device in the treatment of chronic wounds. The study aims to compare the outcomes of standard of care alone versus standard of care combined with plasma treatment.

60 eligible participants presenting with chronic wounds (such as venous leg ulcers or diabetic foot ulcers) will be randomized into two groups:

* One group will receive standard wound care as per clinical practice.
* The other group will receive standard wound care along with cold plasma therapy administered using the Plasana One® device.

  6 participants suffering from pressure ulcers will also be included for an ancillary study.

The study includes both hospital-based and home-based components. Key study procedures include wound assessment through photography, clinical data collection using an electronic case report form (eCRF), and evaluation of patient-reported outcomes such as quality of life (Wound-QoL questionnaire).

Treatments and follow-up visits will be conducted by hospital investigators and home healthcare professionals, depending on the participant's care pathway. Plasma treatment will be delivered by trained nurses during home visits, with gas supplies and device management coordinated by a home care service provider (PSAD).

The primary objective is to evaluate the efficacy of the cold plasma device Plasana One® in the local management of chronic wounds in participants suffering from diabetic foot ulcers and venous leg ulcers, at Week 6.

Secondary objectives include wound healing progression, quality of life, safety of plasma application, and user satisfaction over a 20-week period.

The objective of the ancillary study will be to describe the healing process in pressure ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, age ≥ 18 years,
* Patients affiliated with a social security system or benefiting from such a system,
* Patients able and willing to provide written informed consent,
* Patients able and willing to attend regular follow-up visits during up to 20 weeks, and comply with study procedures,
* Patients whose home healthcare professional is willing to follow the clinical investigation protocol,
* Patient with gas conformed stockage area (ventilated or at least 7m²)
* Patients without infection, or with a local controlled infection,
* Patients with VLU:

  * Patients with wound anteriority between 1 to 12 months
  * Patients with VLU or mixed ulcer of predominantly venous origin (measured ankle brachial index (ABI) such as 1.3 ≥ ABI ≥ 0.8)
  * Patients with VLU between 4 to 30 cm² in surface area,
  * Patients with only one VLU,
  * Patients who have not shown wound healing improvement after wearing compression system for at least two weeks
* Patients with DFU:

  * Patients with wound duration between 1 to 12 months
  * Patients with DFU and with measured ABI ≥ 0.8 or Toe Brachial Index (TBI) ≥ 0.7
  * Patients with DFU between 1 to 30 cm² in surface area,
  * Patients with only one DFU, not between toes,
  * Patients who have not shown wound healing improvement after wearing an offloading system for at least two weeks,
* Patient with PU:

  * Patient with wound duration between 1 to 12 months
  * Patient with PU stage 2 or 3 NPUAP grade,
  * Patient with PU and with ABPI ≥ 0.8 and ≤ 1.3 and/or Toe Brachial Index (TBI) ≥ 0.7 if PU on the foot
  * Patient with PU between 4 to 30 cm² in surface area,
  * Patient with only one PU
  * Patient able and willing to wear off loading system or to be install on pressure relieving system et changing position regularly,

Exclusion Criteria:

* Patients with any other wound treatments other than SOC, Patients who has undergone surgery or surgical revascularization (vascular reconstruction or angioplasty) since less than three months, except for VLU patients who have undergone local graft surgery included in VLU SOC.
* Patients with an active Charcot's neuro-arthropathy as determined by clinical and/or radiographic examination,
* Patients with critical limb ischemia or severe PAD (ankle pressure < 50 mmHg or Toe pressure < 30 mmHg).
* Patients with conditions that may affect wound healing, such as rheumatoid arthritis, scleroderma, or tumor wounds.
* Patients with progressive neoplastic lesions treated by radiotherapy, chemotherapy, hormone therapy or immunosuppressant,
* Patients with non-controlled systemic infection by a suitable antibiotic,
* Patients with suspicion of severe malnutrition,
* Pregnancy or breastfeeding woman, or susceptible to be pregnant,
* Patients with known allergy or hypersensitivity to components of the cold plasma device or standard wound care products,
* Patients included in another study,
* Patients under guardianship or protection of vulnerable adult.
* Patients with implantable electro-medical devices.
* Patients with a history of hypersensitivity or known allergy to medical argon or any component of the device.
* Infected wounds requiring urgent medical or surgical treatment before the application of any device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with Relative Wound Area Reduction (RWAR) ≥ 50% at week 6 from baseline, compared between intervention group and control group, for each indication, measured using digital planimetry software (Pixacare, CE Marked) | From enrollment to week 6.
  The percentage of patients with Relative Wound Area Reduction (RWAR) ≥ 50% at week 6 from baseline, compared between intervention group and control group, for each indication.
  With :
  RWAR; in % : [(SD0 - SW6)/SD0] x 100 SW6 : wound area at week 6 SD0 : wound area at D0
  The wound area will be measured in a standardized way using digital planimetry with Pixacare software, guaranteeing a reproducible and objective measurement.

SECONDARY OUTCOMES:
In each arm, the percentage of patients with Relative Wound Area Reduction (RWAR)≥ 50% at each week from baseline, measured using digital planimetry software (Pixacare, CE Marked) | Each week from baseline to week 20.
  With :
  RWAR; in % : [(SD0 - SW6)/SD0] x 100 SW6 : wound area at week 6 SD0 : wound area at D0
  The wound area will be measured in a standardized way using digital planimetry with Pixacare software, guaranteeing a reproducible and objective measurement.
Time to 100% re-epithelialization in the two patient groups | From baseline to week 20.
  100% re-epithelialization will be assessed by the home healthcare provider or the investigational center of the patient, and confirmed by two other blinded investigators.
The percentage of wounds achieving complete closure defined by 100% re-epithelization, at W6, W12, W20, in both patient groups | At week 6, at week 12 and week 20 post inclusion.
  100% re-epithelialization will be assessed by the home healthcare provider or the investigational center of the patient, and confirmed by two other blinded investigators.
In the two patient groups, the measurement of wound surface from baseline to W6, W12, W20, measured using digital planimetry software (Pixacare, CE Marked) | At week 6, at week 12 and week 20 post inclusion.
In each arm, the number of care procedures (SOC only or SOC + CAP) will be compared between the distinct time points | From baseline to week 20.

OTHER OUTCOMES:
The occurrence and seriousness of adverse events related to the use of Plasana One® | From baseline to week 20.
Score change from baseline based on the Wound-QOL-17 at week 6, at week 12 and week 20 | At week 6, at week 12 and week 20 post inclusion.
Treatment pain evolution based on an Visual Analog Scale | From baseline to week 20.
Usability questionnaire completed at the end of the treatment period by the investigators and nurses, as final users of the device | Week 20
Ancillary outcome for Pressure Ulcers patients only: In the two patient groups, the measurement of wound surface from baseline to W6, W12, W20, measured using digital planimetry software (Pixacare, CE Marked) | From baseline to week 20.
  In each arm for PU patients, the measurement of wound surface from baseline to W6, W12, W20, measured using digital planimetry software (Pixacare, CE Marked)
  As for the primary endpoint, the wound area will be measured in a standardized way using Pixacare software, guaranteeing a reproducible and objective measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Dured Dardari, MD, PhD, Principal Investigator — Centre Hospitalier Sud Francilien

IPD SHARING:
Plan to Share IPD: Undecided